CLINICAL TRIAL: NCT00497770
Title: Non-small Cell Lung Cancer: The Impact of Ethnic Origin on Patients Being Treated Second Line With Pemetrexed - An Observational Study
Brief Title: An Observational Study of the Ethnic Impact of Patients Undergoing Second (2nd) Line Treatment for Non-Small Cell Lung Cancer Using Pemetrexed
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 10733; H3E-US-B001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Caucasian: Caucasian patients receiving Alimta for 2nd line NSCLC
  Interventions: Drug: Pemetrexed
- African American: African American patients receiving Alimta for 2nd line NSCLC
  Interventions: Drug: Pemetrexed
- Asian American: Asian American patients receiving Alimta for 2nd line NSCLC
  Interventions: Drug: Pemetrexed
- Hispanic: Hispanic patients receiving Alimta for 2nd line NSCLC
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Treatment pattern and treatment initiation or changes are solely at the discretion of the physician and the patient
  Other Names: LY231514; Alimta

SUMMARY:
This large, non-randomized observational study is being conducted to provide data about the impact of ethnic origin on outcomes and resource utilization during the 2nd line treatment of non-small cell lung cancer (NSCLC) in a routine medical care setting.

DETAILED DESCRIPTION:
This is a large 1000 patient single arm observational study being conducted to determine the impact of ethnic origin (Caucasian, African-Americans, Asian-Americans, and Hispanics) on patients being treated for 2nd line advanced NSCLC with pemetrexed given in routine clinical practice. Data will be collected on disease control rate by pemetrexed as defined by Response Rate (RR) (Complete Response (CR) + Partial Response (PR)), Stable Disease (SD) and toxicities. In addition, overall survival, progression-free survival, treatment toxicities, activities of daily living, symptom burden and resource utilization will also be observed. To meet the study goals, a total of 400 Caucasians, 200 African- Americans, 200 Asian-Americans, and 200 Hispanics will be accrued to this study.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) (any histologic type)
* Stage IIIB or IV disease
* Should have had 1 line of chemotherapy for Metastatic disease
* Adequate hematologic, hepatic and renal function
* Measurable or evaluable disease

Exclusion Criteria:

* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving pemetrexed for second (2nd) line treatment of non-small cell lung cancer (NSCLC): 400 Caucasians, 200 African-Americans, 200 Asian-Americans, and 200 Hispanic patients will be accrued to this study.
Sampling Method: Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2007-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- United States (37):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campbell, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daly City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poway, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Jose, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunnyvale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greeley, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stamford, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Weston, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kealakekua, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corpus Christi, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galveston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richardson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monroe, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target goals for recruitment were not met due to slow enrollment.
Groups:
- Caucasian: Caucasian participants receiving pemetrexed for second (2nd) line non-small cell lung cancer (NSCLC)
- African American: African American participants receiving pemetrexed for 2nd line NSCLC
- Asian American: Asian American participants receiving pemetrexed for 2nd line NSCLC
- Hispanic: Hispanic participants receiving pemetrexed for 2nd line NSCLC
Period: Overall Study
Arm/Group | Caucasian | African American | Asian American | Hispanic
Started | 304 | 65 | 37 | 28
Completed | 304 | 65 | 37 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caucasian | African American | Asian American | Hispanic | Total
Number analyzed (Participants) | 304 | 65 | 37 | 28 | 434
Age Continuous [Mean (Standard Deviation); unit: years] | 65.64 (9.94) | 62.74 (8.93) | 65.05 (11.31) | 63.14 (13.29) | 64.99 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 22 | 20 | 14 | 199
  Male | 161 | 43 | 17 | 14 | 235
Region of Enrollment [Number; unit: participants]
  United States | 304 | 65 | 37 | 28 | 434
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIB - the cancer has spread to nearby tissue or spread to far away lymph nodes (locally advanced).
  Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver (metastatic).
  participants
    IIIB | 60 | 14 | 8 | 8 | 90
    IV | 244 | 51 | 29 | 20 | 344
Histology of tumor [Number; unit: participants] — This was an observational study, as such, the investigators followed the label recommendations and any changes to the label which occurred during the study, including but not limited to the tumor type.
  participants
    Adenocarcinoma | 191 | 44 | 33 | 25 | 293
    Squamous Cell | 77 | 13 | 2 | 2 | 94
    Other [not adenocarcinoma or squamous cell] | 36 | 8 | 2 | 1 | 47
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 58 | 15 | 12 | 8 | 93
    1 - Ambulatory, Restricted Strenuous Activity | 166 | 39 | 15 | 14 | 234
    2 - Ambulatory, No Work Activities | 53 | 7 | 3 | 2 | 65
    3 - Partially Confined to Bed, Limited Self Care | 8 | 1 | 1 | 1 | 11
    Not available | 19 | 3 | 6 | 3 | 31
Smoking Status [Number; unit: participants]
  Current | 83 | 21 | 0 | 3 | 107
  Former | 196 | 42 | 13 | 18 | 269
  Never | 21 | 2 | 24 | 7 | 54
  Not Collected | 1 | 0 | 0 | 0 | 1
  Unknown | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Disease Control Response (Disease Control Rate)
Description: Disease Control Rate [DCR] is the percentage of participants with Complete Response (CR), Partial Response (PR), Stable Disease (SD), and SD or Incomplete Response (SI). Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=20% increase in sum of longest diameter of target lesions; SD=small changes not meeting above criteria; SI=persistence of 1 or more non-target lesion(s) and/or maintenance of tumor marker level above normal limits.
Time Frame: baseline to measured progressive disease (up to 20 cycles [14 months])
Population: Of the 434 participants enrolled, 50 participants had a response status at the end of pemetrexed treatment indicating "Not done/Missing" and were not included in this analysis.
Measure: Number; unit: percentage of participants
Groups:
- Caucasian: Caucasian participants receiving pemetrexed for 2nd line NSCLC
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 268 | 60 | 30 | 26
percentage of participants | 43.7 | 45.0 | 53.33 | 34.6
Statistical Analysis 1: Comparison: Caucasian vs African American; Test type: Non-Inferiority or Equivalence — A pre-specified logistic regression was used to assess non-inferiority of DCR in African American participants compared with Caucasian participants. The DCR for African Americans was to be considered non-inferior to the DCR for Caucasians if the upper bound of the confidence interval (CI) of the odds ratio (OR) for African American versus Caucasian was <1.78 which corresponds to a difference in proportions of approximately 14% assuming the DCR in the reference group to be 50%; Regression, Logistic — Adjusted:baseline characteristics, income, marital/insurance status, comorbid, time between end of 1st line therapy and start of pemetrexed, prior platinum- or Paclitaxel-containing regimen, number of cycles and best response during 1st line therapy; Odds Ratio (OR) = 0.821, 95% CI 2-sided [0.427 to 1.580]

2. Secondary Outcome: Overall Survival
Description: Overall survival is the duration (months) from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
months | 6.77 (0.38) [5.68 to 7.92] | 6.90 (1.34) [4.53 to 8.94] | 16.0 (1.06) [5.75 to 16.0] | 5.35 (0.91) [2.04 to 12.0]

3. Secondary Outcome: Progression Free Survival
Description: Time from start of second line therapy until death, disease progression, or last contact expressed in months. Participants lost to follow-up (that were alive at last contact) were treated as censored using Kaplan-Meier survival analysis method.
Time Frame: baseline to measured progressive disease or death (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
months | 2.66 [2.40 to 3.35] | 2.99 [2.33 to 4.73] | 5.08 [2.50 to 11.1] | 2.20 [1.81 to 3.71]

4. Secondary Outcome: Functional Status Based on Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to Plan and Prepare Meals
Description: The daily activities assessed: ability to plan and prepare meals. OARS-IADL assesses the participant's ability to plan and prepare meals at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 63.2 | 63.1 | 70.3 | 71.4
  Some Help-baseline | 24.3 | 23.1 | 13.5 | 10.7
  Unable-baseline | 4.9 | 9.2 | 10.8 | 17.9
  Not Done (missing)-baseline | 7.6 | 4.6 | 5.4 | 0.0
  Without Help-end of treatment | 25.3 | 26.2 | 37.8 | 14.3
  Some Help-end of treatment | 9.5 | 13.8 | 8.1 | 10.7
  Unable-end of treatment | 4.3 | 9.2 | 0.0 | 3.6
  Not Done (missing)-end of treatment | 60.9 | 50.8 | 54.1 | 71.4

5. Secondary Outcome: Functional Status Based on the Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to Drive or Use Public Transportation
Description: The daily activities assessed: ability to drive or use public transportation. OARS-IADL assesses the participant's ability to drive or use public transportation at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 62.2 | 63.1 | 62.2 | 50.0
  Some Help-baseline | 29.6 | 32.3 | 29.7 | 50.0
  Unable-baseline | 0.7 | 0.0 | 2.7 | 0.0
  Not Done (missing)-baseline | 7.6 | 4.6 | 5.4 | 0.0
  Without Help-end of treatment | 23.4 | 29.2 | 45.9 | 21.4
  Some Help-end of treatment | 14.8 | 20.0 | 0.0 | 7.1
  Unable-end of treatment | 1.0 | 0.0 | 0.0 | 0.0
  Not Done (missing)-end of treatment | 60.9 | 50.8 | 54.1 | 71.4

6. Secondary Outcome: Functional Status Based on the Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to Handle Personal Finances
Description: The daily activities assessed: ability to handle personal finances. OARS-IADL assesses the participant's ability to handle personal finances at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 78.6 | 67.7 | 83.8 | 71.4
  Some Help-baseline | 11.5 | 26.2 | 8.1 | 17.9
  Unable-baseline | 2.3 | 0.0 | 2.7 | 10.7
  Not Done (missing)-baseline | 7.6 | 6.2 | 5.4 | 0.0
  Without Help-end of treatment | 31.9 | 38.5 | 45.9 | 25.0
  Some Help-end of treatment | 5.6 | 10.8 | 0.0 | 3.6
  Unable-end of treatment | 1.3 | 0.0 | 0.0 | 0.0
  Not Done (missing)-end of treatment | 61.2 | 50.8 | 54.1 | 71.4

7. Secondary Outcome: Functional Status Based on the Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to Perform Housework Activities
Description: The daily activities assessed: ability to perform housework activities. OARS-IADL assesses the participant's ability to perform housework activities at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 44.1 | 44.6 | 54.1 | 42.9
  Some Help-baseline | 38.2 | 33.8 | 32.4 | 32.1
  Unable-baseline | 9.5 | 16.9 | 8.1 | 25.0
  Not Done (missing)-baseline | 8.2 | 4.6 | 5.4 | 0.0
  Without Help-end of treatment | 15.8 | 21.5 | 27.0 | 10.7
  Some Help-end of treatment | 15.5 | 18.5 | 16.2 | 14.3
  Unable-end of treatment | 7.2 | 9.2 | 2.7 | 3.6
  Not Done (missing)-end of treatment | 61.5 | 50.8 | 54.1 | 71.4

8. Secondary Outcome: Functional Status Based on the Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to Prepare and Take Medications
Description: The daily activities assessed: ability to prepare and take medications. OARS-IADL assesses the participant's ability to prepare and take medications at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 79.3 | 73.8 | 86.5 | 85.7
  Some Help-baseline | 12.8 | 21.5 | 5.4 | 7.1
  Unable-baseline | 0.7 | 0.0 | 2.7 | 7.1
  Not Done (missing)-baseline | 7.2 | 4.6 | 5.4 | 0.0
  Without Help-end of treatment | 30.9 | 36.9 | 45.9 | 25.0
  Some Help-end of treatment | 7.6 | 10.8 | 0.0 | 0.0
  Unable-end of treatment | 0.7 | 1.5 | 0.0 | 3.6
  Not Done (missing)-end of treatment | 7.2 | 4.6 | 5.4 | 0.0

9. Secondary Outcome: Functional Status Based on the Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to do the Act of Shopping
Description: The daily activities assessed: ability to do the act of shopping. OARS-IADL assesses the participant's ability to do the act of shopping at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 57.2 | 58.5 | 59.5 | 50.0
  Some Help-baseline | 29.9 | 32.3 | 29.7 | 35.7
  Unable-baseline | 5.6 | 4.6 | 5.4 | 14.3
  Not Done (missing)-baseline | 7.2 | 4.6 | 5.4 | 0.0
  Without Help-end of treatment | 20.1 | 24.6 | 40.5 | 14.3
  Some Help-end of treatment | 14.1 | 21.5 | 5.4 | 14.3
  Unable-end of treatment | 4.6 | 3.1 | 0.0 | 0.0
  Not Done (missing)-end of treatment | 61.2 | 50.8 | 54.1 | 71.4

10. Secondary Outcome: Functional Status Based on the Older Americans Resources and Services Instrumental Activities of Daily Living Scale(OARS-IADL), Ability to Operate the Telephone
Description: The daily activities assessed: ability to operate the telephone. OARS-IADL assesses the participant's ability to operate the telephone at baseline and end of treatment. Responses: ability to do the activity without help, some help, unable, or not done (missing). The percent of participants responding in the different levels of functional ability are provided.
Time Frame: beginning and at end of pemetrexed treatment (up to 20 cycles [14 months])
Population: All participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 304 | 65 | 37 | 28
percentage of participants
  Without Help-baseline | 86.5 | 90.8 | 86.5 | 92.9
  Some Help-baseline | 5.6 | 4.6 | 5.4 | 3.6
  Unable-baseline | 0.0 | 0.0 | 2.7 | 0.0
  Not Done (missing)-baseline | 7.9 | 4.6 | 5.4 | 3.6
  Without Help-end of treatment | 34.9 | 41.5 | 45.9 | 25.0
  Some Help-end of treatment | 3.0 | 7.7 | 0.0 | 3.6
  Unable-end of treatment | 1.3 | 0.0 | 0.0 | 0.0
  Not Done (missing)-end of treatment | 60.9 | 50.8 | 54.1 | 71.4

11. Secondary Outcome: Symptom Score Associated With Treatment as Measured by the M.D. Anderson Symptom Inventory - LC(MDASI-LC)
Description: The symptom score assessed: pain, fatigue, nausea, sleep, distress, shortness of breath, memory, appetite, drowsy, dry mouth, sadness, vomiting, numbness, cough, constipation, general activity, mood, work, relationships with other people, walking, enjoyment. Scores for each item range from 0 to 10, where 0 equaled no symptoms and 10 equaled worst possible symptoms. Assessed at baseline and end of treatment.
Time Frame: Baseline and end of treatment (up to 20 cycles [14 months])
Population: The number of participants who had measurements for the subscale at those time points.
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Caucasian | African American | Asian American | Hispanic
Number analyzed (Participants) | 282 | 65 | 35 | 28
participants
  Pain-baseline (n=281, 62, 35, 28) | 3.37 (3.27) | 3.73 (3.63) | 3.89 (3.32) | 3.75 (3.95)
  Pain-end of treatment (EOT) (n=118, 31, 17, 8) | 3.52 (3.25) | 5.16 (3.69) | 1.82 (2.30) | 1.88 (2.17)
  Fatigue-baseline (n=279, 62, 35, 28) | 4.63 (2.83) | 4.58 (3.11) | 4.14 (2.37) | 5.04 (3.28)
  Fatigue-EOT (n=119, 32, 17, 8) | 4.98 (2.72) | 4.91 (3.30) | 3.71 (2.76) | 4.00 (3.74)
  Nausea-baseline (n=280, 62, 35, 28) | 1.39 (2.54) | 1.55 (2.60) | 1.34 (2.18) | 2.43 (3.49)
  Nausea-EOT (n=118, 30, 17, 8) | 1.76 (2.67) | 1.67 (2.66) | 1.18 (1.33) | 0.75 (1.39)
  Sleep-baseline (n=280, 62, 34, 28) | 3.24 (3.07) | 3.66 (3.59) | 3.21 (3.27) | 4.11 (2.97)
  Sleep-EOT (n=118, 31, 17, 8) | 3.58 (2.97) | 4.16 (3.40) | 2.94 (3.27) | 3.13 (3.80)
  Distress (Upset)-baseline (n=277, 62, 34, 28) | 2.89 (3.01) | 3.00 (3.23) | 2.76 (2.71) | 4.07 (3.57)
  Distress (Upset)-EOT (n=119, 32, 17, 8) | 3.05 (2.94) | 3.22 (3.58) | 2.41 (1.97) | 3.63 (4.10)
  Shortness of Breath-baseline (n=282, 61, 35, 28) | 3.58 (3.06) | 3.70 (3.12) | 2.69 (3.00) | 4.29 (3.40)
  Shortness of Breath-EOT (n=118, 32, 17, 8) | 3.76 (3.12) | 5.06 (3.32) | 1.82 (2.53) | 2.88 (3.44)
  Memory-baseline (n=278, 62, 35, 28) | 2.40 (2.56) | 2.71 (2.56) | 2.09 (2.31) | 2.50 (2.77)
  Memory-EOT (n=119, 32, 17, 8) | 2.47 (2.56) | 2.81 (3.06) | 1.82 (2.38) | 0.63 (1.19)
  Appetite-baseline (n=281, 62, 35, 28) | 2.84 (3.02) | 3.11 (3.38) | 3.37 (2.73) | 4.86 (3.30)
  Appetite-EOT (n=119, 32, 16, 8) | 2.87 (3.01) | 4.72 (4.03) | 2.38 (2.58) | 4.00 (3.74)
  Drowsy-baseline (n=280, 65, 32, 28) | 3.20 (2.79) | 3.32 (2.97) | 2.63 (2.38) | 4.36 (3.18)
  Drowsy-EOT (n=119, 32, 17, 8) | 3.30 (2.84) | 3.69 (3.56) | 1.59 (1.84) | 3.13 (3.18)
  Dry Mouth-baseline (n=279, 62, 35, 28) | 2.89 (2.98) | 2.73 (3.06) | 3.29 (3.19) | 3.36 (3.41)
  Dry Mouth-EOT (n=119, 32, 17, 8) | 2.91 (2.99) | 2.44 (3.04) | 2.71 (2.78) | 2.25 (2.96)
  Sadness-baseline (n=278, 61, 35, 28) | 2.40 (2.81) | 2.57 (3.23) | 2.74 (2.81) | 4.32 (3.51)
  Sadness-EOT (n=119, 32, 17, 8) | 2.39 (2.83) | 2.81 (3.59) | 2.06 (2.08) | 3.88 (3.72)
  Vomiting-baseline (n=282, 62, 35, 28) | 0.74 (1.85) | 0.97 (2.06) | 0.66 (1.35) | 1.25 (2.59)
  Vomiting-EOT (n=119, 32, 17, 8) | 0.97 (1.49) | 1.06 (2.03) | 0.88 (2.03) | 0.13 (0.35)
  Numbness-baseline (n=280, 61, 33, 28) | 2.42 (2.99) | 3.34 (3.26) | 2.76 (2.72) | 2.39 (3.40)
  Numbness-EOT (n=119, 32, 17, 8) | 2.34 (2.64) | 3.84 (3.47) | 2.47 (2.15) | 0.63 (1.77)
  Cough-baseline (n=281, 61, 35, 28) | 2.89 (2.92) | 2.98 (2.91) | 2.63 (2.77) | 2.61 (3.44)
  Cough-EOT (n=119, 31, 16, 8) | 2.50 (2.63) | 3.94 (3.21) | 1.63 (1.96) | 3.13 (3.60)
  Constipation-baseline (n=281, 62 34, 28) | 2.47 (3.11) | 2.37 (3.17) | 2.79 (3.22) | 3.54 (3.86)
  Constipation-EOT (n=119, 32 17, 8) | 2.55 (2.85) | 2.88 (3.50) | 2.47 (3.10) | 1.50 (1.77)
  General Activity-baseline (n=280, 62, 35, 28) | 3.71 (3.13) | 3.56 (3.38) | 2.46 (2.69) | 4.46 (3.89)
  General Activity-EOT (n=119,32,16,8) | 3.89 (3.04) | 4.53 (3.65) | 2.88 (2.70) | 3.63 (3.50)
  Mood-baseline (n=279, 61, 34, 28) | 2.85 (2.96) | 3.11 (3.07) | 2.44 (2.78) | 3.86 (3.76)
  Mood-EOT (n=119, 32, 16, 8) | 2.07 (2.24) | 1.88 (2.23) | 1.89 (2.26) | 1.86 (2.97)
  Work-baseline (n=278, 62, 35, 28) | 3.72 (3.32) | 4.23 (3.86) | 2.51 (2.45) | 4.86 (3.95)
  Work-EOT (n=118, 32, 16, 8) | 4.05 (3.47) | 4.63 (3.72) | 2.81 (2.48) | 4.25 (3.77)
  Relationships with Others-baseline(n=282,61,35,28) | 1.83 (2.53) | 2.41 (3.07) | 2.00 (2.52) | 3.07 (3.57)
  Relationships with Others-EOT (n=118, 31, 16, 8) | 2.17 (2.76) | 2.71 (3.13) | 1.50 (2.31) | 2.75 (3.96)
  Walking-baseline (n=280, 62, 35, 28) | 3.84 (3.15) | 4.00 (3.39) | 2.80 (2.75) | 4.21 (3.35)
  Walking-EOT (n=119, 32, 16, 8) | 4.12 (3.32) | 4.44 (3.56) | 2.94 (2.54) | 4.00 (3.82)
  Enjoyment-baseline (n=282, 61, 35, 28) | 3.33 (3.26) | 3.51 (3.38) | 2.83 (2.81) | 4.39 (4.04)
  Enjoyment-EOT (n=119, 32, 16, 8) | 3.39 (3.16) | 4.00 (3.77) | 2.81 (2.54) | 4.00 (4.75)

ADVERSE EVENTS:
Arm/Group | Caucasian | African American | Asian American | Hispanic
Serious Adverse Events (participants affected / at risk) | 21/304 | 4/65 | 1/37 | 1/28
Other Adverse Events (participants affected / at risk) | 256/304 | 54/65 | 27/37 | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caucasian (N=304) | African American (N=65) | Asian American (N=37) | Hispanic (N=28)
Neutropenia (Blood and lymphatic system disorders) | 8 (10) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (12) | 3 (3) | 1 (1) | 0 (0)
Mucositis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caucasian (N=304) | African American (N=65) | Asian American (N=37) | Hispanic (N=28)
Neutropenia (Blood and lymphatic system disorders) | 55 (76) | 9 (13) | 2 (3) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 55 (84) | 6 (10) | 2 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 45 (59) | 5 (6) | 2 (2) | 2 (4)
Fatigue (General disorders) | 242 (516) | 52 (108) | 27 (57) | 21 (37)
Mucositis (General disorders) | 22 (25) | 9 (12) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 55 (79) | 5 (7) | 2 (3) | 3 (6)

LIMITATIONS AND CAVEATS:
This is an observational study, as such, the investigators followed the label recommendations and any changes to the label which occurred during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days